CLINICAL TRIAL: NCT01502358
Title: A Phase 1 Study To Evaluate The Safety, Tolerability, and Immunogenicity of a Tetravalent Dengue (Serotype 1, 2, 3, and 4) Plasmid DNA Vaccine (TVDV) Formulated With and Without Vaxfectin®
Brief Title: Evaluation of the Safety and the Ability of a DNA Vaccine to Protect Against Dengue Disease
Acronym: TVDV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Vical (Industry); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-11-0007; WRAIR #1839 (Other: WRAIR); NMRC 2011.0012 (Other: NMRC); A-16892 (Other: IRB)
Record Dates: First submitted 2011-12-15; First posted 2011-12-30 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2015-04

CONDITIONS: Dengue Disease; Dengue Fever
Keywords: dengue; dengue fever; dengue disease; tetravalent dengue vaccine; Vaxfectin®
MeSH Terms: conditions — Dengue | interventions — Dengue Vaccines; vaxfectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tetravalent Dengue Vaccine (TVDV) (Experimental): low dose (no adjuvant)
  Interventions: Biological: Tetravalent Dengue Vaccine (TVDV)
- Tetravalent Dengue Vaccine (TVDV) with Vaxfectin® (low-dose) (Experimental): low dose (with adjuvant)
  Interventions: Biological: Tetravalent Dengue Vaccine (TVDV) with Vaxfectin® (low-dose)
- Tetravalent dengue Vaccine (TVDV) with Vaxfectin® (high-dose) (Experimental): high dose (with adjuvant)
  Interventions: Biological: Tetravalent Dengue Vaccine TVDV with Vaxfectin® (High Dose)

INTERVENTIONS:
Biological: Tetravalent Dengue Vaccine (TVDV) — Low dose delivered intramuscularly on Study Days 0, 30 and 90
  Arms: Tetravalent Dengue Vaccine (TVDV)
Biological: Tetravalent Dengue Vaccine (TVDV) with Vaxfectin® (low-dose) — Low dose: TVDV formulated with Vaxfectin®; 1.0 mL volume delivered intramuscularly on Study Days 0, 30 and 90
  Arms: Tetravalent Dengue Vaccine (TVDV) with Vaxfectin® (low-dose)
Biological: Tetravalent Dengue Vaccine TVDV with Vaxfectin® (High Dose) — High dose: TVDV formulated with Vaxfectin®; 1.0 mL volume delivered intramuscularly on Study Days 0, 30 and 90
  Arms: Tetravalent dengue Vaccine (TVDV) with Vaxfectin® (high-dose)

SUMMARY:
The purpose of this study is to determine whether a new investigational dengue vaccine is safe, well-tolerated, and to see if an immune response against dengue disease will be generated.

DETAILED DESCRIPTION:
Arguably the need for a tetravalent dengue vaccine that will effectively induce immunity against all four dengue serotypes has never been greater. Currently, several different approaches are being taken to develop a protective tetravalent dengue vaccine. These include live-attenuated vaccines derived by serial passage in tissue culture, live chimeric vaccines, recombinant protein vaccines and DNA vaccines. While live attenuated and live chimeric vaccines have shown promise in clinical trials, viral competition with suspected immune interference resulting in imbalanced immune responses and reactogenicity with the occurrence of dengue like symptoms remains a concern. It is imperative that any candidate vaccine produce solid immunity against each of the four dengue virus serotypes. Failure to do so may place the recipient of the vaccine at risk for developing severe dengue disease (dengue hemorrhagic fever/dengue shock syndrome) following exposure to the virus serotype to which there was incomplete protective immunity, resulting in antibody dependent enhancement due to the presence of non-neutralizing anti-dengue antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 50 (inclusive) years old at the time of enrollment
* Have negative anti-dengue, Japanese encephalitis, West Nile, and yellow fever ELISA serological tests
* Be informed of the nature of the study and provide written informed consent
* If the subject is of child-producing potential, he/she agrees to practice adequate birth control or abstain from sex
* Have access to the WRAIR Clinical Trials for at least 270 days, and be willing to refrain from participation in other investigational clinical trials
* Be in good general health

Exclusion Criteria-Subjects meeting any of the following criteria will be excluded from the study:

* History of Flavivirus infection or history of Flavivirus vaccine (experimental or licensed product) including Japanese encephalitis, yellow fever, and dengue
* Have a known or suspected hypersensitivity or adverse reaction to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain
* Have received a live-attenuated vaccine within 42 days prior to the initial injection on Day 0 or a subunit or killed vaccine within 30 days of the initial injection on Day 0
* Have a positive screen for hepatitis B surface antigen (HBsAg), hepatitis C antibody, or HIV antibody
* Are pregnant or breastfeeding
* Have donated or received blood, blood products, or plasma within 30 days prior to Day 0
* Have any acute illness, including an oral body temperature >100.4°F, within 7 days before the initial injection on Day 0
* Have a past or current history of malignant disease except for adequately treated skin cancer
* Exclusions include but are not limited to conditions pertaining to or evidence of immunodeficiency; allergies requiring treatment with antigen injections; autoimmune disease; severe migraine headaches; unstable asthma; clinically significant cardiac arrhythmias, diabetes mellitus, thyroid disease, a bleeding disorder or a seizure disorder.
* Have participated in an investigational drug, vaccine, or device study within a period of 30 days prior to Day 0;
* History of splenectomy
* Planned travel to dengue endemic areas during the study period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) or serious adverse events (SAEs) | Up to Day 360
  All AEs and SAEs will be recorded during the entire duration of the study, or up to 360 days.

SECONDARY OUTCOMES:
Percent of subjects (in each group) achieving tetravalent ELISA IgM seroconversion | Days 0-360
  From date of first vaccine dose until seroconversion is achieved, up to 360 days.
Percent of subjects (in each group) achieving tetravalent seroconversion, by dengue plaque reduction MN50 titer | Days 0-360
  From date of first vaccine dose until seroconversion is achieved, up to 360 days.
MN50 titer 1 month (Study Day 120) and Study Days 180 and 270 after vaccine regimen is complete | Following completion of study days 120 and 180 and 270 days after vaccine regimen is complete

CONTACTS AND LOCATIONS:
Overall Officials: Janine R Danko, MD, Principal Investigator — Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research and Clinical Trial Center (WRAIR CTC), Silver Spring, Maryland, United States